CLINICAL TRIAL: NCT00378898
Title: DUAL BRAVO PH MONITORING: A Feasibility Trial
Brief Title: Feasibility of Placing Bravo PH Capsule in Proximal Esophagus
Acronym: bravo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Michael Vaezi, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 060724
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Drug Implants

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- EGD with proximal BRAVO capsule (Active Comparator): Subjects have a second BRAVO capsule placed 10cm proximal to prior BRAVO capsule placement. Fluoroscopy is used to confirm detachment of the monitor 7 days after investigational deployment.
  Interventions: Device: BRAVO capsule; Procedure: Fluoroscopy
- EGD with sham BRAVO capsule placement (Sham Comparator): Subjects have a EGD with BRAVO delivery introducer positioned 10cm proximal to prior BRAVO capsule placement with no BRAVO placed.
  Interventions: Other: sham BRAVO capsule placement

INTERVENTIONS:
Device: BRAVO capsule
  Arms: EGD with proximal BRAVO capsule
Procedure: Fluoroscopy — one time "xray" to determine evacuation of bravo
  Other Names: one time "xray" to determine evacuation of bravo
  Arms: EGD with proximal BRAVO capsule
Other: sham BRAVO capsule placement
  Arms: EGD with sham BRAVO capsule placement

SUMMARY:
Assessing the feasibility and patient tolerance to placement of Bravo PH capsule in proximal esophagus.

There will be no difference in patient-perception of a proximally-placed Bravo esophageal pH monitor compared with a distal monitor.

DETAILED DESCRIPTION:
24-hour pH monitoring is often considered the "gold standard" in the diagnosis of GERD and is increasingly utilized in patients with extra-esophageal symptoms (1). However, the clinical utility of pH monitoring in this patient population remains controversial. An important limitation of traditional pH catheters is their suboptimal sensitivity especially in patients with extraesophageal GERD. Vaezi et al. tested reproducibility and reliability of the proximal and distal esophageal pH probe in 32 patients (2). Among these patients,11 were controls, 10 had distal reflux, and 11 had both proximal and distal reflux. In this group of patients the sensitivity of distal and proximal pH probes were 70% and 55%, respectively. Additionally, a more recent study by Shaker et al. showed the number and duration of hypopharyngeal reflux events to be similar between the control subjects and patients with reflux laryngitis and vasomotor rhinitis (3).

Poor sensitivity of catheter based pH monitoring in detecting acid reflux may be due to day to day variability of test, its less than adequate reliability as well as possible intermittent nature of the reflux events (not recorded in only a 24-hour period) (4). Additionally, since the traditional ambulatory device is commonly placed transnasally through the oropharynx into the esophagus, patients often complain of throat and nose discomfort and usually restrict their daily activity. This potentially leads to false negative findings and reduced test sensitivity. Furthermore, incorrect results may be collected if the pH electrode slips away from the initial manometrically determined placement site. In light of these limitations, a new wireless (catheter free) pH monitoring device was developed to improve patient comfort and increase test sensitivity. The Bravo pH monitoring system (Medtronic Inc, Minneapolis, MN) uses a radiotelemetric capsule temporarily attached to the esophageal mucosa which transmits pH data to a receiver carried on patient's belt.

Although well studied in the distal esophagus, there are currently no studies in adults assessing the feasibility and patient tolerance to placement of this device more proximally. Such a placement may increase the sensitivity of the test and add to our ability to study potential predictors of treatment response in patients with extraesophageal GERD.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will include the following:
* Patients greater than or equal to 18 years of age
* Patients having regularly scheduled upper endoscopy with planned Bravo pH monitor testing
* Patients with known GERD based on symptoms (heartburn, regurgitation) and response to a proton pump inhibitor or esophagitis on EGD as well as those with extraesophageal GERD (cough, asthma and throat discomfort).

Exclusion Criteria:

* Exclusion criteria will include the following:
* Previous surgical procedures to the upper esophagus
* History of bleeding diathesis or coagulopathy
* Stroke or transient ischemic attack within the past 6 months
* GI bleeding within the previous 6 months
* Known esophageal varices
* Significant medical illness (i.e., congestive heart failure)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-09; Primary Completion 2009-03 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael F Vaezi, MD, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- The Vanderbilt Clinic/ Endoscopy Lab, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were 18 years of age or older and scheduled for esophagogastroduodenoscopy (EGD) and wireless pH testing for physiologic assessment of esophageal acid exposure for typical gastroesophageal reflux disease (GERD) symptoms such as heartburn and regurgitation or for extra-esophageal reflux symptoms such as cough or asthma at Vanderbilt.
Groups:
- EGD With BRAVO Capsule: Bravo PH capsule:egd with bravo placement
  Fluoroscopy: one time "xray" to determine evacuation of bravo
Period: Overall Study
Arm/Group | EGD With BRAVO Capsule | EGD With Sham BRAVO Capsule Placement
Started | 22 | 17
Completed | 11 | 11
Not Completed | 11 | 6
Not completed — Withdrawal by Subject | 10 | 5
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: Analysis is based on participants that completed the study
Groups:
- EGD With BRAVO Capsule: Bravo PH capsule: egd with bravo placement
  Fluoroscopy: one time "xray" to determine evacuation of bravo
- Total: Total of all reporting groups
Arm/Group | EGD With BRAVO Capsule | EGD With Sham BRAVO Capsule Placement | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Median (Full Range); unit: years] | 51 [30 to 77] | 50 [19 to 66] | 51 [19 to 77]
Sex/Gender, Customized [Number; unit: participants] — based on participants that completed the study
  participants
    Female | 4 | 5 | 9
    Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants] — based on participants that completed the study
  participants
    United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Patients Requiring Endoscopic Removal of BRAVO Because of Reported Discomfort
Time Frame: 48 hours
Measure: Number; unit: participants
Groups:
- Sham Comparator: EGD With Sham BRAVO Capsule Placement: Subjects have a EGD with BRAVO delivery introducer positioned 10cm proximal to prior BRAVO capsule placement with no BRAVO placed.
Arm/Group | EGD With BRAVO Capsule | Sham Comparator: EGD With Sham BRAVO Capsule Placement
Number analyzed (Participants) | 11 | 11
participants | 2 | 0

2. Secondary Outcome: Subjects Reporting Chest Pain
Description: Edmonton Symptom Assessment is used to measure the presence and change in symptoms.
Time Frame: 48 hours
Population: 2 subjects had to have the BRAVO removed before 48 hours due to reported discomfort in the BRAVO placement group so chest pain scores were obtained for 9 of the 11 subjects.
Measure: Count of Participants; unit: Participants
Groups:
- EGD With Proximal BRAVO Capsule: Subjects have a second BRAVO capsule placed 10cm proximal to prior BRAVO capsule placement. Fluoroscopy is used to confirm detachment of the monitor 7 days after investigational deployment.
  BRAVO capsule
  Fluoroscopy: one time "xray" to determine evacuation of bravo
- EGD With Sham BRAVO Capsule Placement: Subjects have a EGD with BRAVO delivery introducer positioned 10cm proximal to prior BRAVO capsule placement with no BRAVO placed.
  sham BRAVO capsule placement
Arm/Group | EGD With Proximal BRAVO Capsule | EGD With Sham BRAVO Capsule Placement
Number analyzed (Participants) | 9 | 11
Participants | 6 | 3
Statistical Analysis 1: Comparison: EGD With Proximal BRAVO Capsule vs EGD With Sham BRAVO Capsule Placement; Test type: Superiority; p = .047, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Patients underwent baseline EGD and 48-hour wireless pH monitoring. Assessment of symptoms and any adverse events were completed 48 hours after the study intervention.
Groups:
- EGD With BRAVO Capsule: Bravo PH capsule: egd with bravo placement. Analysis is for participants who completed the study.
  Fluoroscopy: one time "xray" to determine evacuation of bravo
- EGS With Sham BRAVO Capsule Placement: Subjects have a EGD with BRAVO delivery introducer positioned 10cm proximal to prior BRAVO capsule placement with no BRAVO placed. Analysis is for participants who completed the study.
Arm/Group | EGD With BRAVO Capsule | EGS With Sham BRAVO Capsule Placement
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 7/11 | 3/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EGD With BRAVO Capsule (N=11) | EGS With Sham BRAVO Capsule Placement (N=11)
Chest pain (Surgical and medical procedures) | 7 | 3 — Increase in baseline symptom score specific to chest pain when compared to visit 3 (48-hr post intervention)

LIMITATIONS AND CAVEATS:
Selection bias may have been a limitation, as patients volunteering may have had worse symptoms and potentially altered esophageal sensitivity as compared to those who opted not to participate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes